CLINICAL TRIAL: NCT07304609
Title: Effects of Lego® Serious Play® for Teach the Trauma Informed Care on the Trauma Informed Care Knowledge, Self Confidence and Satisfaction on Nursing Students
Brief Title: "Effect of LEGO® Serious Play® Trauma-Informed Care Training on Nursing Students
Acronym: Nursing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Tutku KIRÇI TEMİZ, Research Assistant, PhD, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AnkaraMedipolU-SBF-TKT-01
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Nursing
Keywords: trauma informed care; nursing; student; education; Serious Play

STUDY DESIGN:
Intervention Model Description: LEGO® SERIOUS PLAY, education
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LEGO® Serious Play (Experimental): One week after participants received a one-hour theoretical standard training, trauma-informed care was applied using the LEGO® Serious Play® method. Participants learn trauma-informed care principles and different developmental stages in a hands-on way by designing hospital models with LEGO® bricks. Unlike traditional teaching methods, this approach aims to enhance participants' creativity, engagement, and learning motivation.
  Interventions: Other: LEGO® Serious Play®
- Standard Training (No Intervention): Participants received only a one-hour theoretical standard training about trauma-informed care.

INTERVENTIONS:
Other: LEGO® Serious Play® — Participants learn trauma-informed care principles and different developmental stages in a hands-on way by designing hospital models with LEGO® bricks. Unlike traditional teaching methods, this approach aims to enhance participants' creativity, engagement, and learning motivation."
  Arms: LEGO® Serious Play

SUMMARY:
Hospitalization can have traumatic effects on children and their families, highlighting the importance of trauma-informed care in pediatric nursing. Post-hospitalization trauma, anxiety, and depression are frequently observed in both children and parents, negatively affecting health outcomes and treatment adherence. Since trauma-informed care requires a child- and family-centered, safe, and sensitive approach, educating nursing students on this topic is essential. However, this training is often insufficient in nursing curricula, and its abstract and emotionally challenging nature may hinder students' learning. In this context, the LEGO® Serious Play® method, which helps concretize abstract experiences and supports interactive learning, may serve as an effective educational tool. This study aims to evaluate the effects of trauma-informed pediatric care education delivered through the LSP method on nursing students' knowledge, self-confidence, and satisfaction.

DETAILED DESCRIPTION:
Hospitalization is a stressful and traumatic experience for children and their families. Although most children recover physically after hospitalization, many develop psychological problems such as depression, anxiety, and post-traumatic stress. Recent studies indicate that traumatic experiences related to childhood hospitalization are highly prevalent and influence long-term health outcomes. In the systematic review conducted by Stanzel and Sierau (2021), it was found that 13% of pediatric patients exhibited symptoms consistent with post-traumatic stress disorder and 6-8% showed symptoms of depression or anxiety following hospitalization and medical procedures. In the study by Tang et al. (2025), the prevalence of post-traumatic stress in children after hospitalization ranged between 13% and 84.6%, with medical procedures, child-related factors, and the family environment identified as risk factors.

Hospitalization negatively affects treatment adherence in children due to pediatric medical traumatic stress and also leaves traumatic effects on parents. In the study by Terp and Sjöström (2017), it was determined that parents vividly remembered their child's hospitalization even two years later and continued to experience strong feelings of helplessness and fear. The study emphasized that parents who witnessed their child's struggle for life experienced more severe trauma, which led to post-traumatic stress symptoms. In the study by Stremler et al. (2017), 24% of parents of hospitalized children experienced severe anxiety, 51% experienced major depression, and 26% had significant difficulties in decision-making.

The traumatic effects of illness and hospitalization on children and their families have led to increased emphasis on "trauma-informed pediatric care" in pediatric nursing. Trauma-informed pediatric care is based on assessing trauma in every clinical encounter with children and their families. This approach is defined as recognizing the widespread effects of trauma on individuals, identifying trauma symptoms in patients, families, healthcare professionals, and others within the system, integrating this knowledge into policies, procedures, and practices, and preventing re-traumatization. Trauma-informed care is a comprehensive approach grounded in principles of safety, transparency and trustworthiness, peer support, collaboration, empowerment, and cultural sensitivity. Given the profound effects of trauma on children and families, it is essential for pediatric nurses to adopt and implement a trauma-informed pediatric care approach that centers on the trauma experienced by the child and family, the emotional support they need, and their specific needs.

Healthcare professionals should improve their knowledge, attitudes, and skills regarding trauma-informed care. One way to achieve this is through the integration of trauma-informed pediatric care into pediatric nursing curricula. However, most nursing programs do not systematically incorporate this training into their curricula. Furthermore, because trauma-informed care often involves abstract and emotionally intense concepts, it may lead to resistance, avoidance, or superficial learning among students. Therefore, it is important to use interactive and innovative methods in the teaching process that support students' emotional safety and facilitate the expression of their thoughts. One such method is LEGO® SERIOUS PLAY® (LSP).

LEGO® SERIOUS PLAY® (LSP) is a facilitation method initially designed for strategic planning and development and later applied in various fields such as education and research. This method involves participants building models with LEGO® bricks under the guidance of a facilitator, using these models to externalize abstract ideas and experiences, and then sharing the stories of their models with the group. The process typically begins with warm-up activities, followed by participants creating individual models, sharing their stories, and collaboratively developing shared meanings through group models. In this respect, LSP is an effective pedagogical tool that promotes reflective thinking, supports creative exploration, and enables participants to develop new perspectives based on their own knowledge and experiences.

The literature indicates that LSP is a suitable method for the education of nursing students who frequently encounter complex clinical situations. This method has been reported to increase knowledge levels, enhance analytical and reflective thinking skills, promote resilience, and improve self-confidence. In the study conducted by Hayes and Graham (2019) with nursing students, LSP was found to help students think deeply and clearly interpret their learning journey. In the study by McCusker (2019), the use of metaphors such as LSP in education was found to help overcome cultural and traditional barriers, foster understanding and appreciation, and allow for interaction among different ideas and perspectives.

There is no study in the literature in which trauma-informed pediatric nursing care has been taught to nursing students using the LSP method. This study aims to evaluate the effects of trauma-informed pediatric care taught using the LSP method on the knowledge, self-confidence, and satisfaction levels of nursing students taking a pediatric nursing course. By doing so, it seeks to address an important gap in the literature by demonstrating the effectiveness of the LSP method in teaching trauma-informed pediatric care in nursing education.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being enrolled in the Turkish program of the Nursing Department, Faculty of Health Sciences, Ankara Medipol University
* Taking the Pediatric Health and Diseases Nursing course in the Fall semester of the 2025-2026 academic year

Exclusion Criteria:

* Not volunteering to participate in the study
* Being unable to actively participate in the implementation process
* Incomplete completion of data collection instruments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-12-11 (Estimated); Primary Completion 2025-12-25 (Actual); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
TIC Provider Survey | 2 weeks
  This form based on research findings on post-traumatic stress following traumatic medical events in children. The survey consists of 38 items and includes five categories: 1) knowledge about trauma-informed pediatric care (11 items); 2) attitudes and beliefs about trauma-informed pediatric care (6 items); 3) self-efficacy (10 items); 4) trauma-informed care practices (7 items); and 5) perceived barriers to implementing trauma-informed care (4 items). Items assessing knowledge, attitudes, self-efficacy, and perceived barriers were evaluated using 3- or 4-point Likert-type scales appropriate to each category; for example, potential barriers were rated as "not a barrier," "somewhat a barrier," or "significant barrier." Cronbach's alpha values were found to be in the moderate to excellent range for knowledge (0.66), attitude. Higher score indicates a higher level of trauma-informed care knowledge.
Student Satisfaction and Self-Confidence in Learning Scale | 2 weeks
  This scales Cronbach's alpha value was found to be 0.94 for the satisfaction subscale and 0.87 for the self-confidence subscale. The scale consists of two subscales: "Satisfaction with Current Learning" (5 items) and "Self-Confidence in Learning" (7 items), with items rated on a 5-point Likert scale. The total score is obtained by summing the responses to each item of the scale and dividing by the number of items. The minimum score is 1 and the maximum score is 5. A higher score indicates greater satisfaction and higher self-confidence.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Medipol University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data sharing carries the potential to compromise the privacy of participants; therefore, due to ethical responsibility, only anonymized and aggregate data will be published.

REFERENCES:
- [Background] Unver V, Basak T, Watts P, Gaioso V, Moss J, Tastan S, Iyigun E, Tosun N. The reliability and validity of three questionnaires: The Student Satisfaction and Self-Confidence in Learning Scale, Simulation Design Scale, and Educational Practices Questionnaire. Contemp Nurse. 2017 Feb;53(1):60-74. doi: 10.1080/10376178.2017.1282319. Epub 2017 Feb 10. PMID 28084900
- [Background] 26. Jeffries PR, Rizzolo MA. Designing and implementing models for the innovative use of simulation to teach nursing care of ill adults and children: a national, multi-site, multi-method study. New York, NY: National League for Nursing; 2006.
- [Background] Kassam-Adams N, Rzucidlo S, Campbell M, Good G, Bonifacio E, Slouf K, Schneider S, McKenna C, Hanson CA, Grather D. Nurses' views and current practice of trauma-informed pediatric nursing care. J Pediatr Nurs. 2015 May-Jun;30(3):478-84. doi: 10.1016/j.pedn.2014.11.008. Epub 2014 Dec 3. PMID 25481863
- [Background] 24. Kocatepe V, Uslu Y, Unver V, Kayış A, Karabacak U, Aksoy ME. Comparison of the effects of the in situ simulation and simulated clinical immersion methods on cancer nursing students' extravasation management: Randomized controlled trial. Izmir Democracy University Health Sciences Journal - IDUHES. 2023;6(2):348-359. doi:10.52538/iduhes.1327570
- [Background] 23. McCusker S. Everybody's monkey is important: LEGO® Serious Play® as a methodology for enabling equality of voice within diverse groups. Int J Res Method Educ. 2019:1-17. doi:10.1080/1743727X.2019.1621831.
- [Background] 22. Hayes C, Graham Y. Understanding the building of professional identities with the LEGO® SERIOUS PLAY® method using situational mapping and analysis. High Educ Ski Work Learn. 2019;10(1):99-112. doi:10.1108/HESWBL-05-2019-0069.
- [Background] 21. Seifert T, Tseng W. Disadvantaged college students in Taiwan. J Coll Stud Dev. 2017;58(3):264-82.
- [Background] Thomas A, Lubarsky S, Durning SJ, Young ME. Knowledge Syntheses in Medical Education: Demystifying Scoping Reviews. Acad Med. 2017 Feb;92(2):161-166. doi: 10.1097/ACM.0000000000001452. PMID 27782918
- [Background] Warburton T, Brown J, Sandars J. The use of LEGO(R) SERIOUS PLAY(R) within nurse education: A scoping review. Nurse Educ Today. 2022 Nov;118:105528. doi: 10.1016/j.nedt.2022.105528. Epub 2022 Sep 2. PMID 36084451
- [Background] Pfeiffer KM, Grabbe L. An approach to trauma-informed education in prelicensure nursing curricula. Nurs Forum. 2022 Jul;57(4):658-664. doi: 10.1111/nuf.12726. Epub 2022 Apr 24. PMID 35462412
- [Background] Cannon LM, Coolidge EM, LeGierse J, Moskowitz Y, Buckley C, Chapin E, Warren M, Kuzma EK. Trauma-informed education: Creating and pilot testing a nursing curriculum on trauma-informed care. Nurse Educ Today. 2020 Feb;85:104256. doi: 10.1016/j.nedt.2019.104256. Epub 2019 Nov 1. PMID 31759240
- [Background] Loutfy A, Elzeiny A, Alkubati SA, El-Monshed AH, Zoromba MA, Van Belkum C, Mohamed FSA. Undergraduate nursing students' perspectives of trauma-informed care in pediatric nursing: A cross-sectional Egyptian study. J Pediatr Nurs. 2025 Jan-Feb;80:e127-e135. doi: 10.1016/j.pedn.2024.12.002. Epub 2024 Dec 13. PMID 39674704
- [Background] Marsac ML, Kassam-Adams N, Hildenbrand AK, Nicholls E, Winston FK, Leff SS, Fein J. Implementing a Trauma-Informed Approach in Pediatric Health Care Networks. JAMA Pediatr. 2016 Jan;170(1):70-7. doi: 10.1001/jamapediatrics.2015.2206. PMID 26571032
- [Background] 14. Aktan N, Kwong J, Robinson M, Porter S, Rawlins L, Dorsen C. Trauma-informed educational practices: An educational innovation for graduate nursing students. OJIN Online J Issues Nurs. 2023;28(1). doi:10.3912/OJIN.Vol28No01Man02.
- [Background] 13. Wassink Stigter R, Kooijmans R, Asselman MW, Offerman ECP, Nelen W, Helmond P. Facilitators and barriers in the implementation of trauma-informed approaches in schools: a scoping review. Sch Ment Health. 2022;14(3). doi:10.1007/s12310-021-09496-w.
- [Background] 12. Piotrowski CC. ACEs and trauma-informed care. In: Merrick MT, Guinn AS, editors. Adverse Childhood Experiences: Using Evidence to Advance Research, Practice, Policy, and Prevention. 1st ed. Cambridge (MA): Academic Press; 2020. p. 307-28. doi:10.1016/B978-0-12-816065-7.00015-X.
- [Background] 11. Substance Abuse and Mental Health Services Administration (SAMHSA). SAMHSA's concept of trauma and guidance for a trauma-informed approach. HHS Publication No. (SMA) 14-4884. Rockville (MD): SAMHSA; 2014.
- [Background] Kazak AE, Kassam-Adams N, Schneider S, Zelikovsky N, Alderfer MA, Rourke M. An integrative model of pediatric medical traumatic stress. J Pediatr Psychol. 2006 May;31(4):343-55. doi: 10.1093/jpepsy/jsj054. Epub 2005 Aug 10. PMID 16093522
- [Background] Stremler R, Haddad S, Pullenayegum E, Parshuram C. Psychological Outcomes in Parents of Critically Ill Hospitalized Children. J Pediatr Nurs. 2017 May-Jun;34:36-43. doi: 10.1016/j.pedn.2017.01.012. Epub 2017 Mar 6. PMID 28274664
- [Background] Terp K, Sjostrom-Strand A. Parents' experiences and the effect on the family two years after their child was admitted to a PICU-An interview study. Intensive Crit Care Nurs. 2017 Dec;43:143-148. doi: 10.1016/j.iccn.2017.06.003. Epub 2017 Jun 26. PMID 28663106
- [Background] Ben-Ari A, Sela Y, Ben-David S, Ankri YLE, Benarroch F, Aloni R. A Cross Sectional Study to Identify Traumatic Stress, Medical Phobia and Non-Adherence to Medical Care among Very Young Pediatric Patients. Int J Environ Res Public Health. 2023 Jan 8;20(2):1122. doi: 10.3390/ijerph20021122. PMID 36673876
- [Background] Tang M, Chui PL, Chong MC, Liu X. Post-traumatic stress disorder in children after discharge from the pediatric intensive care unit: a scoping review. Eur Child Adolesc Psychiatry. 2025 Feb;34(2):483-496. doi: 10.1007/s00787-024-02505-8. Epub 2024 Jun 25. PMID 38916767
- [Background] Stanzel A, Sierau S. Pediatric Medical Traumatic Stress (PMTS) following Surgery in Childhood and Adolescence: a Systematic Review. J Child Adolesc Trauma. 2021 Aug 21;15(3):795-809. doi: 10.1007/s40653-021-00391-9. eCollection 2022 Sep. PMID 35958723
- [Background] Goddard A, Janicek E, Etcher L. Trauma-informed care for the pediatric nurse. J Pediatr Nurs. 2022 Jan-Feb;62:1-9. doi: 10.1016/j.pedn.2021.11.003. Epub 2021 Nov 17. PMID 34798581
- [Background] Cinar Ozbay S, Boztepe H, Kanbay Y. Nursing students' views on trauma-informed pediatric nursing care and family-centered care. Arch Psychiatr Nurs. 2023 Jun;44:107-113. doi: 10.1016/j.apnu.2023.04.012. Epub 2023 May 4. PMID 37197854
- [Background] Daughtrey HR, Ruiz MO, Felix N, Saynina O, Sanders LM, Anand KJS. Incidence of mental health conditions following pediatric hospital admissions: analysis of a national database. Front Pediatr. 2024 Feb 21;12:1344870. doi: 10.3389/fped.2024.1344870. eCollection 2024. PMID 38450296
- [Background] Triantafyllou C, Matziou V. Aggravating factors and assessment tools for Posttraumatic Stress Disorder in children after hospitalization. Psychiatriki. 2019 Jul-Sep;30(3):264-270. doi: 10.22365/jpsych.2019.303.256. PMID 31685457